CLINICAL TRIAL: NCT03828344
Title: A Phase 1 Randomized, Placebo-Controlled, Double-Blind Study of the Safety and Tolerability of a Single Intravenous Infusion of BX-U001, a Human Umbilical Cord Tissue Derived Mesenchymal Stem Cell Product, for Refractory Rheumatoid Arthritis
Brief Title: Safety and Tolerability of a Single Intravenous Infusion of BX-U001 in Refractory Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylx Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BXU001-RA
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; mesenchymal stem cell; autoimmune
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- hUC-MSC treatment (Experimental): BX-U001 (hUC-MSC suspension) will be tested at dose of 0.75 or 1.5×10^6 cells/kg of body weight via a single IV infusion using a blood transfusion kit.
  Interventions: Biological: hUC-MSC suspension
- Placebo control (Placebo Comparator): The control arm will be given placebo which contains the same cell suspension solution but without cells. Placebo will be given the same way as BX-U001 via a single IV infusion using a blood transfusion kit.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: hUC-MSC suspension — Patients will be treated at dose of 0.75×10^6 cells/kg of body weight (Cohort 1) or 1.5×10^6 cells/kg of body weight (Cohort 2) via a single IV infusion using a blood transfusion kit.
  Other Names: BX-U001
  Arms: hUC-MSC treatment
Biological: Placebo — Placebo contains the same cell suspension as BX-U001 but without cells.
  Arms: Placebo control

SUMMARY:
This is a phase 1, randomized, placebo-controlled, double-blind, single-dose, clinical trial examining the safety and biological effects of allogeneic fresh human umbilical cord tissue-derived mesenchymal stem cell product BX-U001, given by intravenous (IV) infusion, to rheumatoid arthritis (RA) patients with moderate to severe disease activity, who are not well controlled by their current treatments. Two doses of BX-U001 will be tested in 16 patients. The subjects will receive a one-time IV infusion of BX-U001 and monitored for 52 weeks.

DETAILED DESCRIPTION:
This is a phase 1, randomized, placebo-controlled, double-blind, single-dose, clinical trial examining the safety and biological effects of allogeneic fresh human umbilical cord tissue-derived mesenchymal stem cell product BX-U001, given by IV infusion, to RA patients with moderate to severe disease activity, who are not well controlled by their current treatments.

Two cohorts of patients will be recruited sequentially, and each cohort includes 8 patients. In each cohort, eligible patients will be randomized to the two treatment arms at the ratio of 3:1 (BX-U001: Placebo). The patients in the first cohort will receive a single infusion of BX-U001 at dose of 0.75×10^6 cells/kg body weight or placebo. In the second cohort, the patients will receive a single infusion of BX-U001 at dose of 1.5×10^6 cells/kg body weight or placebo. After the one-time infusion on Day 1, patients will be monitored for 52 weeks. During the study, besides BX-U001 or placebo infusion, patients will remain treated with their previous conventional synthetic disease modifying anti-rheumatic drugs (csDMARDs) and nonsteroidal anti-inflammatory drugs (NSAIDs) (other than biologics) in the same dosage/way.

At the end of Week 12, the patients will undergo efficacy evaluations to determine their response to treatment using the response rate of American College of Rheumatology 20% improvement criteria (ACR20). For patients who lack response to treatment as defined by not achieving 20% improvement on tender joint count (TJC) and swollen joint count (SJC) at Week 12, they will receive standard of care treatment including csDMARDs, biologic DMARDs (bDMARDs) and adjunctive agents such as corticosteroids, NSAIDs, and analgesics at Week 14.

The overall study duration is planned to be 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 70, inclusive.
2. Have a diagnosis of RA in agreement with the 2010 ACR classification criteria: Sum of score equal or more than 6/10 in categories A-D including: A, Joint involvement; B, Serology; C, Acute-phase reactant; D, Duration of symptoms.
3. Have established RA > 6 months of symptoms
4. Have had an inadequate response or documented intolerance to available RA therapies including csDMARDs and TNFi bDMARDs.
5. Current use of csDMARD treatment for RA with at least one of the following: methotrexate (up to 25 mg daily), sulfasalazine (up to 3 g daily), hydroxychloroquine (up to 400mg daily), or leflunomide (up to 20mg daily), or any combination of these agents (with the exception of methotrexate and leflunomide) for at least 3 months, with a stable dose (including route of administration for methotrexate) for at least 6 weeks prior to the screening visit (Visit 0)
6. Have SJC of 4 or more out of 28 at screening and baseline
7. Have TJC of 4 or more out of 28 at screening and baseline
8. CRP greater than upper limit of normal (ULN)
9. Positive for RF and/or anti-CCP antibodies but without extra-articular disease or functional limitations
10. Clinically stable with no significant changes in health status within 2 weeks prior to randomization
11. Stated willingness to comply with all study procedures and availability for the duration of the study
12. Patients must be informed of the investigational nature of this study and give written informed consent in accordance with the institutional and hospital guidelines.

Exclusion Criteria:

1. Infections of hepatitis B, hepatitis C, active or latent tuberculosis, or positive for human immunodeficiency virus (HIV)1 or HIV2
2. Any history of ongoing, significant infections or recent serious infection, i.e., requiring hospitalization and or IV antimicrobial treatment in the 3 months prior to screening.
3. Any active inflammatory diseases other than RA.
4. Serum aminotransferase (ALT or AST) levels > 2x ULN
5. Inadequate kidney function, defined as an estimated glomerular filtration rate (eGFR) < 45 ml/min/1.73 m2 using Modification of Diet in Renal Disease (MDRD) 4-variable formula
6. Chronic obstructive pulmonary disease or known lung disease except for mild asthma treated with bronchodilators.
7. Any coexistent active major medical diagnosis of clinically significant cardiovascular, neurological psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease), or hematological abnormalities that are likely to interfere with patient compliance or study assessments/procedures in the investigators' opinion
8. History of transient ischemic attack
9. History of cerebrovascular accident (stroke)
10. Clinically significant heart disease (New York Heart Association, class III and class IV).
11. Surgery or trauma within 14 days.
12. Pregnant, breastfeeding, or desire to become pregnant or unwilling to practice birth control during participation in the study and for twelve months after completing the study infusion, unless surgically sterilized or postmenopausal during the study.
13. Washout period less than 6 months for rituximab or less than 4 weeks for other bDMARDs.
14. Corticosteroid usage at a high dose (i.e., IV or IM corticosteroids or use of oral prednisone equivalent >10 mg/day) or not at a stable dose for the treatment of RA or other diseases within 28 days prior to randomization.
15. Known allergies or had a history of allergy to blood products
16. Blood product usage within 50 days (except albumin)
17. Already participating in another interventional clinical trial or participated in another interventional clinical trial within 3 months before screening.
18. Clinical history of malignancy with the exception of adequately treated cervical carcinoma in situ or basal cell carcinomas.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-20 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AE) and Serious Adverse Events (SAE) | 12 months after infusion
  Total number and rate of AEs and SAEs, related and non-related with BX-U001 infusion will be recorded as a measure of tolerability and safety.

SECONDARY OUTCOMES:
Percentage of participants achieving ACR20 from Baseline at Week 12 and Week 24 | 12 weeks and 24 weeks after infusion
  The ACR20 is a composite measure defined as both improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Percentage of participants achieving ACR50 response from Baseline at Week 12 and Week 24 | 12 weeks and 24 weeks after infusion
  The ACR50 is a composite measure defined as both improvement of 50% in the number of tender and number of swollen joints, and a 50% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Percentage of participants achieving ACR70 response from Baseline at Week 12 and Week 24 | 12 weeks and 24 weeks after infusion
  The ACR70 is a composite measure defined as both improvement of 70% in the number of tender and number of swollen joints, and a 70% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Change from Baseline in the disease activity score 28-joint count using C reactive protein (DAS28-CRP) at Week 12 and Week 24 | 12 weeks and 24 weeks after infusion
  The DAS28-CRP is a composite measure of inflammation in Rheumatoid Arthritis and incorporates a tender and swollen joint count, CRP and Patient Global Assessment of Disease Activity expressed in a Gaussian distribution of variables ranging from 0 to 10. A DAS28-CRP score of <3.2 suggests a low level of disease activity, while a score of >5.1 suggests a high level of disease activity.
Change from Baseline in the health assessment questionnaire disability index (HAQ-DI) score at Week 12 and Week 24 | 12 weeks and 24 weeks after infusion
  The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty when performing daily activities. Each question asks on a scale ranging from 0 to 3 if the categories can be performed without any difficulty (scale 0) up to cannot be done at all (scale 3).
Percentage of participants achieving remission by Simplified Disease Activity Index (SDAI) based criteria at Week 12 and Week 24 | 12 weeks and 24 weeks after infusion
  The SDAI is the numerical sum of five outcome parameters: tender joint count and swollen joint count based on a 28-joint assessment, patient global health assessment and physician global health assessment (from 0=best to 10=worst), and C-reactive protein (CRP). SDAI total score= 0 to 86. SDAI <=3.3 indicates disease remission, >3.3 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity.
Change from Baseline of rheumatoid factor at Week 12 and Week 24 | 12 weeks and 24 weeks after infusion
  Rheumatoid factor blood test result.
Change from Baseline of anti-cyclic citrullinated peptide (anti-CCP) at Week 12 and Week 24 | 12 weeks and 24 weeks after infusion
  Anti-CCP blood test result.